CLINICAL TRIAL: NCT01898598
Title: A Randomized, Double-Blind, Placebo-Controlled, Phase II Study to Assess the Efficacy and Safety of Oral Vismodegib for the Treatment of Basal Cell Carcinoma Preceding Excision by Mohs Micrographic Surgery
Brief Title: A Study of Vismodegib With Surgery in Participants With Previously Untreated Basal Cell Carcinoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ML28726
Record Dates: First submitted 2013-07-03; First posted 2013-07-12 (Estimated); Results first posted 2017-05-08 (Actual); Last update posted 2017-05-08 (Actual); Status verified 2017-03

CONDITIONS: Basal Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Basal Cell | interventions — HhAntag691

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Placebo (Placebo Comparator): Participants will receive matching placebo to vismodegib capsule orally once daily for 12 weeks.
  Interventions: Drug: Placebo
- Vismodegib (Experimental): Participants will receive vismodegib 150 milligrams (mg) capsule orally once daily for 12 weeks.
  Interventions: Drug: Vismodegib

INTERVENTIONS:
Drug: Placebo — Participants will receive matching placebo to vismodegib for 12 weeks.
  Arms: Placebo
Drug: Vismodegib — Participants will receive vismodegib 150 mg oral capsule once a day for 12 weeks
  Arms: Vismodegib

SUMMARY:
This randomized, double-blind, placebo-controlled study will assess the efficacy and safety of vismodegib with surgery in participants with basal cell carcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of non-infected, not recurrent, previously untreated basal cell carcinoma
* Free of any significant physical abnormalities (e.g., tattoos) at the target basal cell carcinoma site
* Willing and able to participate in the study as an outpatient and agreement to make frequent visits to the clinic during the treatment and follow-up periods and to comply with study requirements

Exclusion Criteria:

* Prior treatment with vismodegib
* Known hypersensitivity to any of the study drug excipients
* Any metastatic basal cell carcinoma
* Any locally advanced basal cell carcinoma considered to be inoperable or to have a medical contraindication to surgery
* Evidence of clinically significant and unstable diseases or conditions (e.g., cardiovascular, immunosuppressive, hematologic)
* Any dermatological disease at the target basal cell carcinoma site that may cause difficulty with examination
* Recent, current, or planned participation in another experimental drug study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2014-01-23 (Actual); Primary Completion 2016-01-26 (Actual); Study Completion 2016-01-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (21):
- United States (21):
  - Mayo Clinic, Scottsdale, Arizona
  - Moy-Fincher-Chipps Facial Plastics and Dermatology, Beverly Hills, California
  - Scripps Clinic, La Jolla, California
  - Loma Linda University Medical Center, Loma Linda, California
  - Stanford University, Palo Alto, California
  - California Pacific Medical Center, San Francisco, California
  - Univ of Calif-San Francisco, San Francisco, California
  - Spencer Derma & Skin Surg Ctr, St. Petersburg, Florida
  - Northwestern University, Chicago, Illinois
  - Laser & Skin Surgery Center of Indiana, Carmel, Indiana
  - University of Minnesota, Minneapolis, Minnesota
  - Beth Israel Cancer Center; West Campus, New York, New York
  - University of Rochester Medical Center; University Dermatology Associates, Rochester, New York
  - Mariwalla Dermatology, West Islip, New York
  - The Skin Surgery Center, Winston-Salem, North Carolina
  - Oregon Health & Science University; Department of Dermatology, Portland, Oregon
  - Penn State Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - MD Anderson Cancer Center, Houston, Texas
  - Huntsman Cancer Institute at The University of Utah, Salt Lake City, Utah
  - University of Wisconsin, Madison, Wisconsin

RESULTS

PARTICIPANT FLOW:
Groups:
- Vismodegib: Participants received vismodegib 150 milligrams (mg) capsule orally once daily for 12 weeks.
- Placebo: Participants received matching placebo to vismodegib capsule orally once daily for 12 weeks.
Period: Overall Study
Arm/Group | Vismodegib | Placebo
Started | 12 | 6
Treated | 11 | 5
Completed | 8 | 4
Not Completed | 4 | 2
Not completed — Adverse Event | 1 | 0
Not completed — Withdrawal by Subject | 3 | 0
Not completed — Lost to Follow-up | 0 | 1
Not completed — Other | 0 | 1

BASELINE CHARACTERISTICS:
Population: The Intent-to-treat (ITT) population included all randomized participants who received at least one dose of study treatment.
Groups:
- Vismodegib: Participants received vismodegib 150 mg capsule orally once daily for 12 weeks.
- Total: Total of all reporting groups
Arm/Group | Vismodegib | Placebo | Total
Number analyzed (Participants) | 11 | 5 | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 71.5 (10.87) | 73.6 (7.27) | 72.2 (9.68)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2
  Male | 10 | 4 | 14

OUTCOME MEASURES:

1. Primary Outcome: Percent Change in Target Basal Cell Carcinoma (BCC) Expected Surgical Defect Area at Mohs Micrographic Surgery (MMS) Visit
Description: The percent change in target BCC expected surgical defect area was defined as ([baseline expected surgical defect area - expected surgical defect area at MMS visit]/ baseline expected surgical defect area) × 100 percent (%) where expected surgical defect area was manually outlined on a digital photograph and measured by a computer (computer aided planimetry). MMS visit was defined as the visit that occurred within 2 weeks of the last study treatment.
Time Frame: Baseline, MMS visit (Week 12-14)
Population: ITT population. Here 'Number of participants analyzed' represents participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: Percent change in surgical defect area
Arm/Group | Vismodegib | Placebo
Number analyzed (Participants) | 7 | 4
Percent change in surgical defect area | 31.52 (35.580) | 46.30 (20.232)

2. Secondary Outcome: Actual Change in Target BCC Expected Surgical Defect Area at MMS Visit
Description: Actual change was defined as (baseline expected surgical defect area - expected surgical defect area at MMS visit). MMS visit was defined as the visit that occurred within 2 weeks of the last study treatment. Expected surgical defect area was manually outlined on a digital photograph and measured by a computer (computer aided planimetry).
Time Frame: Baseline, MSS Visit (Week 12-14)
Population: ITT Population. Here 'Number of participants analyzed' represents participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: Square millimeter (mm^2)
Arm/Group | Vismodegib | Placebo
Number analyzed (Participants) | 7 | 4
Square millimeter (mm^2) | 70.16 (82.483) | 93.33 (35.768)

3. Secondary Outcome: Percentage Change in Target BCC Actual Tumor-Free Margin Excision Area at MMS Visit
Description: Percent change in target BCC actual tumor-free margin excision area was defined as = (expected surgical defect area pre-treatment - actual tumor-free margin excision area at MMS visit) / expected surgical defect area pre-treatment) * 100%. The actual tumor-free margin excision area (includes 2 millimeters [mm] margin) was measured during MMS. The area was photographed and traced on the digital photograph then calculated by computer-aided planimetry. MMS visit was defined as the visit that occurred within 2 weeks of the last study treatment.
Time Frame: Baseline, MMS visit (Week 12-14)
Population: ITT. Here 'Number of participants analyzed' represents participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: Percent change in margin excision area
Arm/Group | Vismodegib | Placebo
Number analyzed (Participants) | 6 | 4
Percent change in margin excision area | -12.24 (78.775) | 25.29 (65.763)

4. Secondary Outcome: Percentage of Participants With Clinical Response
Description: Clinical response was defined as a complete response (CR) or partial response (PR) at the post-treatment MMS excision. CR was defined as no histological evidence of BCC. PR was defined as a reduction of at least 50 % in the expected surgical defect area with histologic evidence of residual BCC. MMS visit was defined the visit that occurred within 2 weeks of the last study treatment.
Time Frame: MMS visit (Week 12-14)
Population: ITT population.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Vismodegib | Placebo
Number analyzed (Participants) | 11 | 5
Percentage of participants | 18.2 [2.3 to 51.8] | 40.0 [5.3 to 85.3]
Statistical Analysis 1: Comparison: Vismodegib vs Placebo; The 95 % confidence interval (CI) for the difference in response rates was computed using the exact unconditional confidence limits method; Test type: Superiority or Other; Difference in Clinical Response Rates = -21.8, 95% CI 2-sided [-71.6 to 32.1]

5. Secondary Outcome: Percentage of Participants With Skip Area
Description: Skip area was defined as the presence of non-contiguous residual tumor at the MMS visit, as determined by an independent dermatopathologist. MMS visit occurred within 2 weeks of the last study treatment.
Time Frame: MMS visit (Week 12-14)
Population: ITT population.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Vismodegib | Placebo
Number analyzed (Participants) | 11 | 5
Percentage of participants | 0.0 [0.0 to 28.5] | 40.0 [5.3 to 85.3]
Statistical Analysis 1: Comparison: Vismodegib vs Placebo; Test type: Superiority or Other; Percentage Difference = -40.0, 95% CI 2-sided [-85.3 to 14.2]

6. Secondary Outcome: Percentage of Participants With BCC Recurrence
Time Frame: Baseline, 12, 24, and 52 weeks post MMS Visit (MMS Visit = Week 12-14)
Population: This outcome was based on the cumulative data post MMS Visit and due to early study termination with very few enrolled participants, complete data for this outcome measure could not be collected.
Arm/Group | Vismodegib | Placebo
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Baseline up to 52 weeks after last study treatment (Last Study Treatment = Week 12)
Description: Safety population, included all participants who received at least one dose of study treatment.
Arm/Group | Vismodegib | Placebo
Serious Adverse Events (participants affected / at risk) | 3/11 | 0/5
Other Adverse Events (participants affected / at risk) | 9/11 | 2/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Vismodegib (N=11) | Placebo (N=5)
Gastric ulcer (Gastrointestinal disorders) | 1 | 0
Oesophagitis (Gastrointestinal disorders) | 1 | 0
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Vismodegib (N=11) | Placebo (N=5)
Diarrhoea (Gastrointestinal disorders) | 3 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1
Fatigue (General disorders) | 1 | 0
Influenza like illness (General disorders) | 0 | 1
Bronchitis (Infections and infestations) | 1 | 0
Laceration (Injury, poisoning and procedural complications) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 7 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1
Dysgeusia (Nervous system disorders) | 5 | 0
Ageusia (Nervous system disorders) | 1 | 0
Nerve compression (Nervous system disorders) | 1 | 0
Anxiety (Psychiatric disorders) | 0 | 1
Confusional state (Psychiatric disorders) | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 3 | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 1
Hypertension (Vascular disorders) | 1 | 0

LIMITATIONS AND CAVEATS:
The study was discontinued early by the Sponsor and due to a small sample size, no conclusions can be drawn.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.